CLINICAL TRIAL: NCT01380574
Title: Safety of Cardioversion of Acute Atrial Fibrillation
Acronym: FinCV
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Juhani Airaksinen, Professor, Turku University Hospital
Other Study IDs: K23
Record Dates: First submitted 2011-06-16; First posted 2011-06-27 (Estimated); Last update posted 2012-06-28 (Estimated); Status verified 2012-06

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; cardioversion; stroke; thromboembolism
MeSH Terms: conditions — Atrial Fibrillation; Stroke; Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to investigate the complications of cardioversion of acute (<48 hours duration) atrial fibrillation (AF).

Primary Outcome Measures:

- Incidence and predictors of thromboembolic complications, especially stroke, and death <31 days after cardioversion of acute AF

Secondary Outcome Measures:

* Number of therapy non-responder and early recurrence of AF
* Bleeding complications during the 31 days follow-up
* Hemodynamic complications of cardioversion

Estimated Enrollment: 3000 cases

Study Start Date: Jun 2011

Estimated Study Completion Date: December 2011

DETAILED DESCRIPTION:
It has been a common practice to perform cardioversion of acute (<48 hour) AF without any anticoagulation. The new European guidelines recommend that anticoagulation should be started already before cardioversion in all patients with CHADS2VASC score indicating need for long-term oral anticoagulation. The evidence behind these guidelines is, however, scarce. In this retrospective study we collect data on the safety of acute AF cardioversion from emergency rooms of two university hospitals and one secondary referral center from the years 2003-2010.

Inclusion criteria:

All patients admitted to emergency room because of acute AF in whom electrical or pharmacological cardioversion was attempted <48 from the beginning of the symptoms.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to emergency room because of acute AF in whom electrical or pharmacological cardioversion was attempted <48 from the beginning of the symptoms

Exclusion Criteria:

* duration of the AF is unknown or >48 hours

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients admitted to emergency room because of acute AF in whom electrical or pharmacological cardioversion was attempted <48 from the beginning of the symptoms.
Sampling Method: Non-Probability Sample
Enrollment: 7700 (Actual)
Dates: Start 2011-06; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Incidence and predictors of thromboembolic complications, especially stroke, and death <31 days after cardioversion of acute AF | 31 days

SECONDARY OUTCOMES:
Number of therapy non-responder and early recurrence of AF | 31 days
Bleeding complications during the 31 days follow-up | 31 days
Hemodynamic complications of cardioversion | 31 days

CONTACTS AND LOCATIONS:
Overall Officials: Juhani Airaksinen, Professor, Principal Investigator — Turku University Hospital
Locations (3):
- Finland (3):
  - Kuopio University Hospital, Kuopio
  - Satakunta Central Hospital, Pori
  - Turku University Hospital, Turku

REFERENCES:
- [Derived] Jaakkola S, Nuotio I, Hartikainen JEK, Airaksinen KEJ. Early Cardioversion for Acute Atrial Fibrillation in Low Stroke Risk Patients Is Safe Without Anticoagulation. J Am Coll Cardiol. 2020 Jul 14;76(2):226-227. doi: 10.1016/j.jacc.2020.04.076. No abstract available. PMID 32646574
- [Derived] Jaakkola J, Hartikainen JE, Kiviniemi T, Nuotio I, Nammas W, Gronberg T, Karmi A, Ylitalo A, Airaksinen KE. Ventricular rate during acute atrial fibrillation and outcome of electrical cardioversion: The FinCV Study. Ann Med. 2015 Jun;47(4):341-5. doi: 10.3109/07853890.2015.1031821. Epub 2015 May 6. PMID 25943162
- [Derived] Nuotio I, Hartikainen JE, Gronberg T, Biancari F, Airaksinen KE. Time to cardioversion for acute atrial fibrillation and thromboembolic complications. JAMA. 2014 Aug 13;312(6):647-9. doi: 10.1001/jama.2014.3824. No abstract available. PMID 25117135
- [Derived] Airaksinen KE, Gronberg T, Nuotio I, Nikkinen M, Ylitalo A, Biancari F, Hartikainen JE. Thromboembolic complications after cardioversion of acute atrial fibrillation: the FinCV (Finnish CardioVersion) study. J Am Coll Cardiol. 2013 Sep 24;62(13):1187-92. doi: 10.1016/j.jacc.2013.04.089. Epub 2013 Jul 10. PMID 23850908